CLINICAL TRIAL: NCT01126580
Title: The Impact of LY2189265 Versus Metformin on Glycemic Control in Early Type 2 Diabetes Mellitus (AWARD-3: Assessment of Weekly AdministRation of LY2189265 in Diabetes-3)
Brief Title: A Study in Participants With Type 2 Diabetes Mellitus (AWARD-3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11375; H9X-MC-GBDC (Other: Eli Lilly and Company); CTRI/2010/091/003036 (Registry Identifier: Clinical Trials Register India)
Record Dates: First submitted 2010-05-18; First posted 2010-05-19 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; dulaglutide; Injections, Subcutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1.5 mg LY2189265 (Experimental): LY2189265 (Dulaglutide): 1.5 milligrams (mg), subcutaneously (SC), once weekly for 52 weeks
  Placebo: 1 tablet per day, orally, for Week 1; 2 tablets per day, orally, for Week 2; 3 tablets per day, orally, for Week 3; 4 or at least 3 tablets, orally, for Weeks 4 through Week 52
  Interventions: Drug: LY2189265; Drug: Placebo (oral)
- 0.75 mg LY2189265 (Experimental): LY2189265 (Dulaglutide): 0.75 milligrams (mg), subcutaneously (SC), once weekly for 52 weeks
  Placebo: 1 tablet per day, orally, for Week 1; 2 tablets per day, orally, for Week 2; 3 tablets per day, orally, for Week 3; 4 or at least 3 tablets, orally, for Weeks 4 through Week 52
  Interventions: Drug: LY2189265; Drug: Placebo (oral)
- Metformin (Active Comparator): Metformin: 500 milligrams per day (mg/day), orally, for Week 1; 1000 mg/day, orally, for Week 2; 1500 mg/day, orally, for Week 3; 2000 or at least 1500 mg/day, orally, for Weeks 4 through Week 52
  Placebo: subcutaneously (SC), once weekly for 52 weeks
  Interventions: Drug: Metformin; Drug: Placebo (subcutaneous)

INTERVENTIONS:
Drug: Metformin
  Arms: Metformin
Drug: LY2189265
  Other Names: Dulaglutide
  Arms: 0.75 mg LY2189265; 1.5 mg LY2189265
Drug: Placebo (oral)
  Arms: 0.75 mg LY2189265; 1.5 mg LY2189265
Drug: Placebo (subcutaneous)
  Arms: Metformin

SUMMARY:
The purpose of this study is to determine if LY2189265 is safe and effective in reducing glycosylated hemoglobin (HbA1c) as compared to metformin in participants with Type 2 Diabetes.

DETAILED DESCRIPTION:
The term rescue therapy in this trial was defined primarily as additional nontrial antidiabetic medication for the management of severe, persistent hyperglycemia or alternative antidiabetic medication following study drug discontinuation. For efficacy analyses, participants who received rescue medication were included in the analysis population, but only measurements obtained prior to taking rescue therapy were included in the efficacy analysis. For safety analyses, with the exception of hypoglycemia outcomes, all measurements including those obtained after taking rescue therapy were included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes for greater than or equal to 3 months and less than or equal to 5 years based on the disease diagnostic criteria (refer to the World Health Organization's [WHO] Classification of Diabetes).
* Are treatment-naïve, not optimally controlled with diet and exercise alone, or are taking 1 oral antihyperglycemic medication (OAM) as monotherapy (excluding thiazolidinediones). For those on 1 OAM, the dose must be less than or equal to 50% the maximum authorized per local label.
* Are able and willing to tolerate a minimum dose of 1500 milligrams per day (mg/day) or up to 2000 mg/day of metformin.
* Have glycosylated hemoglobin (HbA1c) greater than or equal to 6.5% to less than or equal to 9.5%.
* Females of childbearing potential (not surgically sterilized and between menarche and 1-year postmenopausal) must: a) test negative for pregnancy at screening based on a serum pregnancy test, and b) agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug; or c) not be breastfeeding.
* Have a stable weight (plus or minus 5%) greater than or equal to 3 months prior to screening.
* Have a body mass index (BMI) between 23 and 45 kilograms per square meter (kg/m^2), inclusive.
* Are well-motivated, capable, and willing to: a) perform self-monitored blood glucose (SMBG) testing; b) learn how to self-inject treatment (LY2189265 or placebo) and c) maintain a study diary.

Exclusion Criteria:

* Have type 1 diabetes mellitus.
* Are being or have been treated with any of the following medications: a) chronically treated with insulin for the treatment of diabetes in the past; however, a short-term use of insulin more than 3 months prior to screening is allowable, b) glucagon-like peptide 1 (GLP-1) analogs within 3 months prior to this screening, c) drugs to cause weight loss within 3 months prior to screening, d) thiazolidinediones (TZDs) within 3 months prior to screening, e) chronically treated (greater than or equal to 14 days) with an oral glucocorticoid or have received this type of therapy within 4 weeks prior to screening, or f) illegal drugs.
* Have had 1 or more cases of uncontrolled diabetes that required hospitalization in the 6 months prior to screening.
* Have stomach problems, have chronically taken medication to increase movement in the digestive tract or slow down the emptying of the digestive tract, or have had gastric bypass (bariatric) surgery.
* Have had problems with the heart or brain in the past 2 months prior to screening, such as a heart attack, chest pain, heart failure, heart bypass operation, angioplasty or stent insertion, a heart rhythm problem, or a stroke.
* Have a serum creatinine result which shows a greater than or equal to 1.5 milligrams per deciliter (mg/dL) for men or greater than or equal to 1.4 mg/dL for women.
* Have a problem with the liver or pancreas.
* Have a creatinine clearance result which shows less than 60 milliliters per minute (mL/min), evidence of a significant active, uncontrolled endocrine (hormone), or active autoimmune abnormality.
* Have a serum calcitonin test which shows greater than or equal to 20 picograms per milliliter (pcg/mL) at the time of screening.
* Have a family history of medullary C-cell hyperplasia or endocrine neoplasia type 2A or type 2B.
* Have cancer (except for skin cancer) or have been in remission from cancer for less than 5 years.
* Have had an organ transplant except for corneal transplant.
* Have received treatment within the last 30 days with a drug which has not been regulatory approved.
* Have participated in a medical, surgical, or pharmaceutical study where these types of procedures were performed within 30 days prior to screening.
* Have any condition that is a contraindication to or would interfere with medications provided for this study to treat diabetes.
* Have a blood disorder that would interfere with the drawing of blood glucose measurements or lab samples.
* Have previously participated or signed an informed consent document for this same type of study and study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 807 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (91):
- United States (28):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buena Park, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burbank, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Redlands, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Mateo, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gurnee, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southfield, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eugene, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beaver, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johnstown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Levittown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Georgetown, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olympia, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Selah, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
- Argentina (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Isidro
- Brazil (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fortaleza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halifax, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
- Croatia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dubrovnik
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osijek
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Slavonski Brod
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb
- Czechia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beroun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nový Jičín
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- Finland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nurmijärvi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oulu
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Bouëxière
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mûrs-Erigné
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vieux-Condé
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gebhardshain
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neunkirchen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Potsdam
- India (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chennai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagpur
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampico
- Poland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Puerto Rico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Galati
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reşiţa
- Slovakia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Banská Bystrica
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trebišov
- South Africa (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halfway House
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kempton Park
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Somerset West
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucheon-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Begonte
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Granada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
- United Kingdom (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Penzance, Cornwall
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, County Durham
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Greater London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveleys, Lancashire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Crawley
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nottingham

REFERENCES:
- [Derived] Gnesin F, Thuesen ACB, Kahler LKA, Madsbad S, Hemmingsen B. Metformin monotherapy for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Jun 5;6(6):CD012906. doi: 10.1002/14651858.CD012906.pub2. PMID 32501595
- [Derived] Boustani MA, Pittman I 4th, Yu M, Thieu VT, Varnado OJ, Juneja R. Similar efficacy and safety of once-weekly dulaglutide in patients with type 2 diabetes aged >/=65 and <65 years. Diabetes Obes Metab. 2016 Aug;18(8):820-8. doi: 10.1111/dom.12687. Epub 2016 Jun 7. PMID 27161178
- [Derived] Yu M, Van Brunt K, Varnado OJ, Boye KS. Patient-reported outcome results in patients with type 2 diabetes treated with once-weekly dulaglutide: data from the AWARD phase III clinical trial programme. Diabetes Obes Metab. 2016 Apr;18(4):419-24. doi: 10.1111/dom.12624. Epub 2016 Feb 4. PMID 26691396
- [Derived] Umpierrez G, Tofe Povedano S, Perez Manghi F, Shurzinske L, Pechtner V. Efficacy and safety of dulaglutide monotherapy versus metformin in type 2 diabetes in a randomized controlled trial (AWARD-3). Diabetes Care. 2014 Aug;37(8):2168-76. doi: 10.2337/dc13-2759. Epub 2014 May 19. PMID 24842985

RESULTS

PARTICIPANT FLOW:
Groups:
- 1.5 mg LY2189265: LY2189265 (Dulaglutide): 1.5 milligrams (mg), subcutaneously (SC), once weekly for 52 weeks
  Placebo: orally, twice daily for 52 weeks
- 0.75 mg LY2189265: LY2189265 (Dulaglutide): 0.75 milligrams (mg), subcutaneously (SC), once weekly for 52 weeks
  Placebo: orally, twice daily for 52 weeks
- Metformin: Metformin: 2000 milligrams per day (mg/day) or at least 1500 mg/day, orally, for 52 weeks
  Placebo: subcutaneously (SC), once weekly for 52 weeks
Period: Overall Study
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Started | 269 | 270 | 268
Received at Least 1 Dose of Study Drug | 269 | 270 | 268
Completed 26 Weeks | 233 | 242 | 226
Completed | 220 | 218 | 213
Not Completed | 49 | 52 | 55
Not completed — Adverse Event | 14 | 8 | 12
Not completed — Withdrawal by Subject | 11 | 19 | 14
Not completed — Sponsor Decision | 5 | 4 | 7
Not completed — Physician Decision | 1 | 1 | 2
Not completed — Entry Criteria Not Met | 1 | 1 | 2
Not completed — Lack of Efficacy | 2 | 3 | 4
Not completed — Protocol Violation | 0 | 1 | 2
Not completed — Lost to Follow-up | 15 | 13 | 9
Not completed — Treatment Non-compliance | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of LY2189265 or Metformin.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin | Total
Number analyzed (Participants) | 269 | 270 | 268 | 807
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.51 (10.38) | 55.90 (10.68) | 55.26 (10.10) | 55.56 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 152 | 147 | 454
  Male | 114 | 118 | 121 | 353
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 90 | 87 | 95 | 272
  Not Hispanic or Latino | 179 | 183 | 173 | 535
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 29 | 28 | 28 | 85
  Asian | 21 | 20 | 20 | 61
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 17 | 22 | 14 | 53
  White | 201 | 198 | 201 | 600
  More than one race | 1 | 2 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 77 | 80 | 74 | 231
  Slovakia | 8 | 9 | 9 | 26
  Finland | 3 | 5 | 4 | 12
  Spain | 12 | 11 | 12 | 35
  United Kingdom | 0 | 1 | 1 | 2
  India | 9 | 11 | 9 | 29
  France | 12 | 12 | 13 | 37
  Czech Republic | 10 | 9 | 8 | 27
  Mexico | 24 | 25 | 23 | 72
  Canada | 10 | 9 | 11 | 30
  Puerto Rico | 14 | 10 | 15 | 39
  Argentina | 27 | 27 | 26 | 80
  Poland | 7 | 6 | 5 | 18
  Brazil | 2 | 2 | 3 | 7
  Croatia | 3 | 4 | 4 | 11
  Romania | 14 | 13 | 13 | 40
  South Africa | 12 | 11 | 12 | 35
  Germany | 22 | 21 | 21 | 64
  Korea, Republic of | 3 | 4 | 5 | 12
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 92.67 (18.79) | 91.79 (18.67) | 92.40 (19.23) | 92.28 (18.87)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m^2) | 33.66 (5.65) | 33.08 (5.84) | 33.05 (5.06) | 33.26 (5.53)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 2.65 (1.50) | 2.60 (2.17) | 2.63 (1.77) | 2.63 (1.83)
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 7.63 (0.92) | 7.58 (0.87) | 7.60 (0.82) | 7.60 (0.87)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 26-week Endpoint in Glycosylated Hemoglobin (HbA1c)
Description: Least Squares (LS) means were calculated using analysis of covariance (ANCOVA) with country, treatment, and prior medication group (previous oral antihyperglycemic medication [OAM] versus no previous OAM) as fixed effects and baseline HbA1c as a covariate.
Time Frame: Baseline, 26 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable HbA1c data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 265 | 265 | 265
percentage of glycosylated hemoglobin | -0.78 (0.06) | -0.71 (0.06) | -0.56 (0.06)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Metformin; The study was designed with 90% power to detect non-inferiority of 1.5 mg LY2189265 vs Metformin on HbA1c change from baseline at the 26-week primary endpoint with a margin of 0.4%, a standard deviation of 1.3%, and a 2-sided alpha of 0.05 assuming no true difference between treatments. This corresponds to 223 participants per arm, with an assumed drop-out rate of 11%; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of 0.4% was used; p < 0.001, ANCOVA — The p-value is adjusted for multiplicity using a tree-gatekeeping strategy. To determine significance, the p-value is compared to the family-wise 1-sided Type I error of 0.025. The confidence interval is not adjusted for multiplicity; LS Mean Difference = -0.22, 95% CI 2-sided [-0.36 to -0.08]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of 0.4% was used; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.15, 95% CI 2-sided [-0.29 to -0.01]
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Metformin; Superiority analysis; Test type: Superiority or Other; p = 0.002, ANCOVA — Tree gatekeeping strategy to control the family-wise Type I error rate was applied; LS Mean Difference = -0.22, 95% CI 2-sided [-0.36 to -0.08]
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Metformin; Superiority analysis; Test type: Superiority or Other; p = 0.020, ANCOVA — Tree gatekeeping strategy to control the family-wise Type I error rate was applied; LS Mean Difference = -0.15, 95% CI 2-sided [-0.29 to -0.01]

2. Secondary Outcome: Change From Baseline to 52-week Endpoint in Glycosylated Hemoglobin (HbA1c)
Description: as for outcome 1
Time Frame: Baseline, 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 265 | 265 | 265
percentage of glycosylated hemoglobin | -0.70 (0.07) | -0.55 (0.07) | -0.51 (0.07)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Metformin; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of 0.4% was used; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.19, 95% CI 2-sided [-0.35 to -0.02]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of 0.4% was used; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.04, 95% CI 2-sided [-0.20 to 0.12]
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Metformin; Superiority analysis; Test type: Superiority or Other; p = 0.024, ANCOVA — Tree gatekeeping strategy to control the family-wise Type I error rate was applied; LS Mean Difference = -0.19, 95% CI 2-sided [-0.35 to -0.02]
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Metformin; Superiority analysis; Test type: Superiority or Other; p = 0.299, ANCOVA — Tree gatekeeping strategy to control the family-wise Type I error rate was applied; LS Mean Difference = -0.04, 95% CI 2-sided [-0.20 to 0.12]

3. Secondary Outcome: Percentage of Participants Achieving a Glycosylated Hemoglobin (HbA1c) of Less Than 7% and Less Than or Equal to 6.5% at 26 and 52 Weeks
Description: The percentage of participants achieving HbA1c level less than 7.0% and less than or equal to 6.5% was analyzed with a logistic regression model with baseline, prior medication group, and treatment as factors included in the model.
Time Frame: 26 weeks and 52 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 265 | 265 | 265
percentage of participants
  HbA1c less than 7%, 26 weeks | 61.5 | 62.6 | 53.6
  HbA1c less than or equal to 6.5%, 26 weeks | 46.0 | 40.0 | 29.8
  HbA1c less than 7%, 52 weeks | 60.0 | 53.2 | 48.3
  HbA1c less than or equal to 6.5%, 52 weeks | 42.3 | 34.7 | 28.3
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.023, Regression, Logistic — Treatment comparison for HbA1c less than 7.0% at 26 weeks
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.021, Regression, Logistic — Treatment comparison for HbA1c less than 7.0% at 26 weeks
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Metformin; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison for HbA1c less than or equal to 6.5% at 26 weeks
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.011, Regression, Logistic — Treatment comparison for HbA1c less than or equal to 6.5% at 26 weeks
Statistical Analysis 5: Comparison: 1.5 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.001, Regression, Logistic — Treatment comparison for HbA1c less than 7% at 52 weeks
Statistical Analysis 6: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.269, Regression, Logistic — Treatment comparison for HbA1c less than 7% at 52 weeks
Statistical Analysis 7: Comparison: 1.5 mg LY2189265 vs Metformin; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison for HbA1c less than or equal to 6.5% at 52 weeks
Statistical Analysis 8: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.134, Regression, Logistic — Treatment comparison for HbA1c less than or equal to 6.5% at 52 weeks

4. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Fasting Blood Glucose
Description: Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, prior medication group, visit, and treatment-by-visit interaction as fixed effects, baseline fasting blood glucose as a covariate, and participant as a random effect.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable fasting blood glucose data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 267 | 265 | 264
millimoles per liter (mmol/L)
  26 weeks (n=244, 247, 245) | -1.61 (0.13) | -1.46 (0.13) | -1.34 (0.13)
  52 weeks (n=207, 210, 194) | -1.56 (0.14) | -1.00 (0.14) | -1.15 (0.14)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.079, Mixed Models Analysis — Treatment comparison at 26 weeks
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.451, Mixed Models Analysis — Treatment comparison at 26 weeks
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis — Treatment comparison at 52 weeks
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.402, Mixed Models Analysis — Treatment comparison at 52 weeks

5. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Daily Mean Blood Glucose Values From the 8-point Self-monitored Blood Glucose (SMBG) Profiles
Description: The SMBG data were collected at the following 8 time points: pre-morning meal; 2 hours post-morning meal; pre-midday meal; 2 hours post-midday meal; pre-evening; 2 hours post-evening meal; bedtime; and 3AM or 5 hours after bedtime. Least Squares (LS) means of the mean of the 8 time points (daily mean) were calculated using analysis of covariance (ANCOVA) with country, treatment, and prior medication group as fixed effects and baseline daily mean as a covariate.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable SMBG data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 211 | 207 | 218
millimoles per liter (mmol/L)
  26 weeks (n=195, 200, 211) | -1.98 (0.15) | -1.75 (0.14) | -1.68 (0.14)
  52 weeks (n=197, 200, 212) | -1.99 (0.16) | -1.71 (0.16) | -1.58 (0.15)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.061, ANCOVA — Treatment comparison at 26 weeks
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.647, ANCOVA — Treatment comparison at 26 weeks
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.022, ANCOVA — Treatment comparison at 52 weeks
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.469, ANCOVA — Treatment comparison at 52 weeks

6. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Body Weight
Description: Least Squares (LS) means were calculated using analysis of covariance (ANCOVA) with country, treatment, and prior medication group as fixed effects and baseline body weight as a covariate.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable body weight data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 269 | 270 | 268
kilograms (kg)
  26 weeks (n=267, 269, 267) | -2.29 (0.24) | -1.36 (0.24) | -2.22 (0.24)
  52 weeks (n=267, 269, 267) | -1.93 (0.29) | -1.09 (0.29) | -2.20 (0.29)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.811, ANCOVA — Treatment comparison at 26 weeks
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.003, ANCOVA — Treatment comparison at 26 weeks
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.440, ANCOVA — Treatment comparison at 52 weeks
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.001, ANCOVA — Treatment comparison at 52 weeks

7. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Body Mass Index (BMI)
Description: Body mass index is an estimate of body fat based on body weight divided by height squared. Least Squares (LS) means were calculated using analysis of covariance (ANCOVA) with country, treatment, and prior medication group as fixed effects and baseline BMI as a covariate.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable BMI data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: kilograms per meter squared (kg/m^2)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 267 | 269 | 267
kilograms per meter squared (kg/m^2)
  26 weeks | -0.86 (0.09) | -0.51 (0.09) | -0.82 (0.09)
  52 weeks | -0.73 (0.11) | -0.42 (0.10) | -0.83 (0.11)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.750, ANCOVA — Treatment comparison at 26 weeks
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.003, ANCOVA — Treatment comparison at 26 weeks
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.412, ANCOVA — Treatment comparison at 52 weeks
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.001, ANCOVA — Treatment comparison at 52 weeks

8. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Homeostasis Model Assessment of Beta-cell Function
Description: The homeostatic model assessment (HOMA) quantifies insulin resistance and beta-cell function. HOMA2-B is a computer model that uses fasting plasma insulin and glucose concentrations to estimate steady-state beta cell function (%B) as a percentage of a normal reference population (normal young adults). HOMA2-S is a computer model that uses fasting plasma insulin and glucose concentrations to estimate insulin sensitivity (%S) as percentages of a normal reference population (normal young adults). The normal reference populations were set at 100%. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, prior medication group, visit, and treatment-by-visit interaction as fixed effects, baseline HOMA2 as a covariate, and participant as a random effect.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable HOMA2-%B or HOMA2-%S data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: percentage of HOMA2
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 245 | 242 | 242
percentage of HOMA2
  HOMA2-%B, 26 weeks (n=207, 207, 215) | 36.55 (3.42) | 28.96 (3.44) | 14.11 (3.37)
  HOMA2-%B, 52 weeks (n=179, 185, 170) | 29.97 (3.46) | 22.5 (3.46) | 9.77 (3.51)
  HOMA2-%S, 26 weeks (n=207, 207, 215) | 0.95 (2.29) | 2.71 (2.29) | 9.99 (2.25)
  HOMA2-%S, 52 weeks (n=179, 185, 170) | 5.29 (2.43) | 1.84 (2.43) | 10.83 (2.48)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Metformin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of HOMA2-%B at 26 weeks
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of HOMA2-%B at 26 weeks
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Metformin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of HOMA2-%B at 52 weeks
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — Treatment comparison of HOMA2-%B at 52 weeks
Statistical Analysis 5: Comparison: 1.5 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — Treatment comparison of HOMA2-%S at 26 weeks
Statistical Analysis 6: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis — Treatment comparison of HOMA2-%S at 26 weeks
Statistical Analysis 7: Comparison: 1.5 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.077, Mixed Models Analysis — Treatment comparison of HOMA2-%S at 52 weeks
Statistical Analysis 8: Comparison: 0.75 mg LY2189265 vs Metformin; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — Treatment comparison of HOMA2-%S at 52 weeks

9. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in the Impact of Weight on Activities of Daily Living (IW-ADL) Score
Description: The Impact of Weight on Activities of Daily Living (renamed the Ability to Perform Physical Activities of Daily Living [APPADL]) questionnaire contains 7 items that assess how difficult it is for participants to engage in certain activities considered to be integral to normal daily life, such as walking, standing and climbing stairs. Items are scored on a 5-point numeric rating scale where 5 = "not at all difficult" and 1 = "unable to do". The individual scores from all 7 items are summed and a single total score is calculated and may range between 7 and 35. A higher score indicates better ability to perform activities of daily living. Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) adjusted by treatment, country, prior medication group, gender, and baseline score.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable APPADL data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 266 | 268 | 266
units on a scale
  26 weeks (n=247, 251, 247) | 0.09 (0.33) | 0.19 (0.32) | 0.02 (0.32)
  52 weeks (n=247, 252, 248) | 0.39 (0.33) | -0.05 (0.33) | 0.28 (0.33)

10. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in the Impact of Weight on Self-Perception (IW-SP) Score
Description: The Impact of Weight on Self-Perception (IW-SP) questionnaire contains 3 items that assess how often the participants' body weight affects how happy they are with their appearance and how often they feel self-conscious when out in public. Items are scored on a 5-point numeric rating scale where 5 = never and 1 = always. A single total score is calculated by summing the scores for all 3 items. Total score ranges between 3 and 15, where a higher score is indicative of better self-perception. Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) adjusted by treatment, country, prior medication group, gender, and baseline score.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable IW-SP data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 268 | 270 | 268
units on a scale
  26 weeks (n=248, 254, 249) | 0.72 (0.19) | 0.63 (0.18) | 0.79 (0.18)
  52 weeks (n=249, 255, 250) | 0.45 (0.19) | 0.61 (0.19) | 0.75 (0.19)

11. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in the Diabetes Treatment Satisfaction Questionnaire (DTSQ) Score, Status Version
Description: The Diabetes Treatment Satisfaction Questionnaire status version (DTSQs) is used to assess participant treatment satisfaction at each study visit. The questionnaire consists of 8 items, 6 of which (1 and 4 through 8) assess treatment satisfaction. Each item is rated on a 7-point Likert scale. Scores from the 6 treatment satisfaction items are summed to a Total Treatment Satisfaction Score, which ranges from 0 (very dissatisfied) to 36 (very satisfied). Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) adjusted by treatment, country, prior medication group, gender, and baseline score.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable DTSQs data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) used to impute missing postbaseline values. If there were no data after randomization, endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 266 | 267 | 267
units on a scale
  26 weeks (n=244, 249, 241) | 1.93 (0.39) | 1.81 (0.38) | 2.04 (0.39)
  52 weeks (n=245, 251, 244) | 1.82 (0.44) | 1.29 (0.43) | 1.94 (0.44)

12. Secondary Outcome: Diabetes Treatment Satisfaction Questionnaire (DTSQ) Score, Change Version
Description: The Diabetes Treatment Satisfaction Questionnaire change (DTSQc) score is used to assess relative change in participant satisfaction from baseline. The questionnaire consists of 8 items, 6 of which (1 and 4 through 8) assess treatment satisfaction. Each item is rated on a 7-point Likert scale. The scores from the 6 treatment satisfaction items are summed to a Total Treatment Satisfaction Score, which ranges from -18 (much less satisfied) to +18 (much more satisfied). Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) adjusted by treatment, country, prior medication group, gender, and baseline score.
Time Frame: 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable DTSQc data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) used to impute missing postbaseline values. If there were no data after randomization, endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 230 | 235 | 230
units on a scale | 12.92 (0.52) | 12.73 (0.50) | 12.58 (0.51)

13. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in the Diabetes Symptoms Checklist Participant-reported Outcome (DSC-r) Score
Description: The Diabetes Symptoms Checklist-revised (DSC-r) was designed to assess the presence and perceived burden of diabetes-related symptoms. Respondents were to consider troublesomeness of 34 symptoms on a 5-point scale ranging from 5="extremely" to 1="not at all." For symptoms/side-effects not experienced, the item was scored as 0. Symptoms were grouped into the following subscales: psychology-fatigue, psychology-cognitive, neurology-pain, neurology-sensory, cardiology, ophthalmology, hypoglycemia, and hyperglycemia. Subscale scores were calculated as the sum of the given subscale divided by the total number of items in the scale. Total score was computed from the sum of the 8 subscales and ranged from 0 to 40. Higher scores indicate greater symptom burden. Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) adjusted by treatment, country, prior medication group, gender, and baseline score.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable DSC-r data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 267 | 270 | 267
units on a scale
  26 weeks (n=245, 253, 248) | 0.24 (0.36) | -0.16 (0.35) | 0.41 (0.35)
  52 weeks (n=247, 255, 249) | 0.49 (0.39) | 0.42 (0.39) | 0.59 (0.39)

14. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events at 26 and 52 Weeks
Description: A treatment-emergent adverse event (TEAE) was defined as an event that first occurs or worsens (increases in severity) after baseline regardless of causality or severity. The number of participants with one or more TEAE is summarized cumulatively at 26 and 52 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: 26 weeks and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 269 | 270 | 268
participants
  26 weeks | 163 | 150 | 151
  52 weeks | 179 | 177 | 170

15. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Electrocardiogram Parameters, Fridericia Corrected QT (QTcF) Interval and PR Interval
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave and was calculated from electrocardiogram (ECG) data using Fridericia's formula: QTc = QT/RR^0.33. Corrected QT (QTc) is the QT interval corrected for heart rate and RR, which is the interval between two R waves. PR is the interval between the P wave and the QRS complex. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, prior medication group, visit, and treatment-by-visit interaction as fixed effects, baseline interval as a covariate, and participant as a random effect.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable ECG QTcF interval or PR interval data.
Measure: Least Squares Mean (Standard Error); unit: milliseconds (msec)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 269 | 270 | 268
milliseconds (msec)
  QTcF interval, 26 weeks (n=230, 237, 221) | 2.60 (1.17) | 1.38 (1.16) | -0.91 (1.18)
  QTcF interval, 52 weeks (n=212, 212, 205) | 3.76 (1.20) | 0.73 (1.19) | -0.53 (1.21)
  PR interval, 26 weeks (n=226, 235, 218) | -0.04 (1.12) | -0.01 (1.10) | -2.04 (1.13)
  PR interval, 52 weeks (n=209, 210, 201) | 1.15 (1.18) | 1.53 (1.17) | -2.88 (1.19)

16. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Electrocardiogram Parameters, Heart Rate
Description: Electrocardiogram (ECG) heart rate was measured. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, prior medication group, visit, and treatment-by-visit interaction as fixed effects and baseline interval as a covariate.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable ECG heart rate data.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 267 | 268 | 264
beats per minute (bpm)
  26 weeks (n=230, 237, 221) | 1.60 (0.60) | 2.57 (0.59) | 0.82 (0.61)
  52 weeks (n=212, 212, 205) | 2.02 (0.66) | 2.36 (0.66) | 1.27 (0.67)

17. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Pulse Rate
Description: Sitting pulse rate was measured. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, prior medication group, visit, and treatment-by-visit interaction as fixed effects, baseline interval as a covariate, and participant as a random effect.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable pulse rate data.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 269 | 270 | 268
beats per minute (bpm)
  26 weeks (n=244, 251, 239) | 2.39 (0.58) | 2.14 (0.57) | 1.59 (0.58)
  52 weeks (n=221, 219, 215) | 1.84 (0.57) | 1.63 (0.57) | 1.12 (0.57)

18. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Blood Pressure
Description: Sitting systolic blood pressure (SBP) and sitting diastolic blood pressure (DBP) were measured. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, prior medication group, visit, and treatment-by-visit interaction as fixed effects, baseline interval as a covariate, and participant as a random effect.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable blood pressure data.
Measure: Least Squares Mean (Standard Error); unit: milliliters of mercury (mmHg)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 269 | 270 | 268
milliliters of mercury (mmHg)
  SBP, 26 weeks (n=244, 251, 239) | -1.89 (0.89) | -2.61 (0.88) | -0.91 (0.89)
  SBP, 52 weeks (n=221, 219, 215) | -0.11 (0.88) | -2.74 (0.88) | -0.98 (0.88)
  DBP, 26 weeks (n=244, 251, 239) | 0.05 (0.57) | -1.02 (0.56) | -0.64 (0.58)
  DBP, 52 weeks (n=221, 219, 215) | 0.31 (0.60) | -1.37 (0.59) | -0.38 (0.60)

19. Secondary Outcome: Percent Change From Baseline to 26 and 52 Weeks in Total Cholesterol
Description: Percent changes in total cholesterol were assessed using analysis of variance (ANOVA) on the rank-transformed data with only treatment included in the model.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable cholesterol data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Median (Inter-Quartile Range); unit: percentage change in total cholesterol
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 258 | 257 | 256
percentage change in total cholesterol
  26 weeks (n=244, 244, 243) | -3.86 [-10.83 to 5.24] | -1.77 [-9.78 to 7.57] | -3.51 [-12.19 to 5.45]
  52 weeks (n=247, 248, 245) | -1.69 [-11.11 to 7.45] | -0.78 [-10.02 to 8.10] | -3.88 [-12.14 to 5.69]

20. Secondary Outcome: Percentage Change From Baseline to 26 and 52 Weeks in High Density Lipoprotein Cholesterol (HDL-C)
Description: Percentage changes in HDL-C were assessed using analysis of variance (ANOVA) on the rank-transformed data with only treatment included in the model.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable HDL-C data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing
Measure: Median (Inter-Quartile Range); unit: percentage change in HDL-C
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 259 | 257 | 257
percentage change in HDL-C
  26 weeks (n=246, 244, 244) | 2.39 [-4.11 to 13.54] | 4.20 [-5.66 to 14.66] | 5.78 [-2.66 to 14.13]
  52 weeks (n=248, 248, 246) | 4.95 [-4.55 to 13.17] | 2.31 [-5.16 to 12.56] | 4.32 [-6.56 to 13.64]

21. Secondary Outcome: Percentage Change From Baseline to 26 and 52 Weeks in Low Density Lipoprotein Cholesterol (LDL-C)
Description: Percentage changes in LDL-C were assessed using analysis of variance (ANOVA) on the rank-transformed data with only treatment included in the model.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable LDL-C data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing
Measure: Median (Inter-Quartile Range); unit: percentage change in LDL-C
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 249 | 249 | 243
percentage change in LDL-C
  26 weeks (n=233, 231, 221) | -6.86 [-18.26 to 8.20] | -2.70 [-15.33 to 9.15] | -8.97 [-20.21 to 5.00]
  52 weeks (n=236, 240, 231) | -2.06 [-15.93 to 9.31] | -2.34 [-15.22 to 10.56] | -7.23 [-18.56 to 4.36]

22. Secondary Outcome: Percentage Change From Baseline to 26 and 52 Weeks in Triglycerides
Description: Percentage changes in triglycerides were assessed using analysis of variance (ANOVA) on the rank-transformed data with only treatment included in the model.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable triglyceride data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing
Measure: Median (Inter-Quartile Range); unit: percentage change in triglycerides
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 266 | 265 | 265
percentage change in triglycerides
  26 weeks (n=252, 252, 253) | -2.35 [-22.32 to 13.61] | -1.96 [-21.66 to 22.63] | 2.56 [-16.00 to 23.79]
  52 weeks (n=255, 256, 254) | -4.27 [-22.91 to 19.23] | -0.86 [-22.31 to 25.37] | 1.91 [-21.65 to 24.04]

23. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Pancreatic Enzymes
Description: Amylase (total and pancreas-derived [PD]) and lipase concentrations were measured.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable pancreatic enzyme data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Median (Inter-Quartile Range); unit: units per liter (U/L)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 266 | 267 | 267
units per liter (U/L)
  Amylase (total), 26 weeks | 7.00 [2.00 to 13.00] | 6.00 [0.00 to 13.00] | 4.00 [-2.00 to 10.00]
  Amylase (total), 52 weeks | 5.50 [-1.00 to 13.00] | 5.00 [-1.00 to 13.00] | 4.00 [-2.00 to 9.00]
  Amylase (PD), 26 weeks | 5.00 [2.00 to 9.00] | 4.00 [1.00 to 7.00] | 1.00 [-1.00 to 5.00]
  Amylase (PD), 52 weeks | 4.00 [1.00 to 7.00] | 3.00 [0.00 to 8.00] | 2.00 [-1.00 to 5.00]
  Lipase, 26 weeks | 7.00 [1.00 to 16.00] | 5.00 [0.00 to 13.00] | 1.00 [-4.00 to 8.00]
  Lipase, 52 weeks | 5.00 [-1.00 to 13.00] | 5.00 [0.00 to 12.00] | 1.00 [-4.00 to 6.00]

24. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Serum Calcitonin
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin with evaluable serum calcitonin data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter (pcg/mL)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 266 | 267 | 267
picograms per milliliter (pcg/mL)
  26 weeks | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  52 weeks | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

25. Secondary Outcome: Number of Participants With Treatment Emergent Anti-LY2189265 Antibodies
Description: A participant was considered to have treatment emergent LY2189265 anti-drug antibodies (ADA) if the participant had at least one titer that was treatment-emergent relative to baseline, defined as a 4-fold or greater increase in titer from baseline measurement. The total number of treatment emergent ADA was not analyzed at 26 weeks.
Time Frame: Baseline through 52 weeks
Population: Participants who received at least one dose of LY2189265 with evaluable LY2189265 ADA data.
Measure: Number; unit: participants
Groups:
- 1.5 mg or 0.75 mg LY2189265: LY2189265 (Dulaglutide): 1.5 milligrams (mg) or 0.75 mg, subcutaneously (SC), once weekly for 52 weeks
  Placebo: orally, twice daily for 52 weeks
Arm/Group | 1.5 mg or 0.75 mg LY2189265
Number analyzed (Participants) | 521
participants | 10

26. Secondary Outcome: Number of Self-reported Hypoglycemic Events at 26 and 52 Weeks
Description: Hypoglycemic events were classified as severe (defined as episodes requiring the assistance of another person to actively administer resuscitative actions), documented symptomatic (defined as any time a participant feels that he/she is experiencing symptoms and/or signs associated with hypoglycemia, and has a plasma glucose level of less than or equal to 70 milligrams per deciliter [mg/dL]), or asymptomatic (defined as events not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose of less than or equal to 70 mg/dL). A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 weeks and 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin. Only pre-rescue measurements were used.
Measure: Number; unit: events
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 269 | 270 | 268
events
  Severe, 26 weeks (n=241, 248, 236) | 0 | 0 | 0
  Severe, 52 weeks (n=214, 217, 199) | 0 | 0 | 0
  Documented Symptomatic, 26 weeks (n=241, 248, 236) | 2 | 6 | 2
  Documented Symptomatic, 52 weeks (n=214, 217, 199) | 7 | 8 | 2
  Asymptomatic, 26 weeks (n=241, 248, 236) | 19 | 9 | 13
  Asymptomatic, 52 weeks (n=214, 217, 199) | 5 | 9 | 9

27. Secondary Outcome: Rate of Self-reported Hypoglycemic Events at 52 Weeks
Description: Hypoglycemic events were classified as severe (defined as episodes requiring the assistance of another person to actively administer resuscitative actions), documented symptomatic (defined as any time a participant feels that he/she is experiencing symptoms and/or signs associated with hypoglycemia, and has a plasma glucose level of less than or equal to 70 milligrams per deciliter [mg/dL]), or asymptomatic (defined as events not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose of less than or equal to 70 mg/dL). The 1-year adjusted rate of hypoglycemic events is summarized cumulatively at 52 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 52 weeks
Population: Participants who received at least one dose of LY2189265 or Metformin. Only pre-rescue measurements were used.
Measure: Mean (Standard Deviation); unit: events per participant per year
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 269 | 270 | 268
events per participant per year
  Severe | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Documented Symptomatic | 0.62 (8.91) | 0.15 (0.72) | 0.09 (0.50)
  Asymptomatic | 0.24 (1.26) | 0.30 (1.85) | 0.18 (0.79)

28. Secondary Outcome: Number of Participants With Adjudicated Pancreatitis at 52 Weeks Plus 30-day Follow up
Description: The number of participants with pancreatitis confirmed by adjudication is summarized cumulatively at 52 weeks plus 30-day follow up. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 52 weeks plus 30-day follow up
Population: Participants who received at least one dose of LY2189265 or Metformin. Only pre-rescue measurements were used.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 269 | 270 | 268
participants | 0 | 0 | 0

29. Secondary Outcome: Number of Participants With Adjudicated Cardiovascular Events at 52 Weeks Plus 30-day Follow up
Description: Information on cardiovascular (CV) risk factors was collected at baseline. Data on any new CV event was prospectively collected using a CV event electronic case report form. Deaths and nonfatal cardiovascular adverse events (AEs) were adjudicated by an external committee of physicians with cardiology expertise. Nonfatal cardiovascular AEs to be adjudicated included myocardial infarction, hospitalization for unstable angina, hospitalization for heart failure, coronary interventions, and cerebrovascular events, including cerebrovascular accident (stroke) and transient ischemic attack. The number of participants with CV events confirmed by adjudication is summarized cumulatively at 52 weeks plus 30-day follow up. Serious and all other non-serious adverse events regardless of causality are summarized in the Reported Adverse Events module.
Time Frame: Baseline through 52 weeks plus 30-day follow up
Population: Participants who received at least one dose of LY2189265 or Metformin.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Number analyzed (Participants) | 269 | 270 | 268
participants
  Any CV Event | 1 | 2 | 1
  Any Fatal CV Event | 0 | 0 | 0
  Any Nonfatal CV Event | 1 | 2 | 1

30. Secondary Outcome: Measurement of LY2189265 Drug Concentration for Pharmacokinetics: Area Under the Concentration Curve (AUC)
Description: Evaluable pharmacokinetic concentrations from the 4-week, 13-week, 26-week, and 52-week timepoints were combined and utilized in a population approach to determine the population mean estimate and standard deviation at steady-state.
Time Frame: 4 weeks, 13 weeks, 26 weeks, and 52 weeks
Population: Participants who received at least one dose of LY2189265 with evaluable LY2189265 concentration data.
Measure: Mean (Standard Deviation); unit: nanogram hours per milliliter (ng*hr/mL)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265
Number analyzed (Participants) | 144 | 146
nanogram hours per milliliter (ng*hr/mL) | 12036 (5385) | 5919 (1548)

ADVERSE EVENTS:
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Metformin
Serious Adverse Events (participants affected / at risk) | 15/269 | 20/270 | 16/268
Other Adverse Events (participants affected / at risk) | 177/269 | 178/270 | 170/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1.5 mg LY2189265 (N=269) | 0.75 mg LY2189265 (N=270) | Metformin (N=268)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 3 (3) | 0 (0)
Paradoxical drug reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Echinococciasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatic echinococciasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/155 (0) | 0/152 (0) | 1/147 (1)
Tongue carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/155 (1) | 0/152 (0) | 0/147 (0)
Bipolar II disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.5 mg LY2189265 (N=269) | 0.75 mg LY2189265 (N=270) | Metformin (N=268)
Abdominal distension (Gastrointestinal disorders) | 13 (18) | 13 (19) | 10 (14)
Abdominal pain (Gastrointestinal disorders) | 11 (16) | 10 (11) | 6 (7)
Constipation (Gastrointestinal disorders) | 18 (23) | 12 (13) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 31 (37) | 26 (30) | 39 (44)
Dyspepsia (Gastrointestinal disorders) | 12 (15) | 8 (22) | 6 (7)
Nausea (Gastrointestinal disorders) | 53 (76) | 31 (45) | 43 (50)
Vomiting (Gastrointestinal disorders) | 26 (32) | 20 (24) | 14 (70)
Bronchitis (Infections and infestations) | 7 (8) | 11 (11) | 9 (9)
Influenza (Infections and infestations) | 9 (11) | 11 (14) | 8 (13)
Nasopharyngitis (Infections and infestations) | 14 (16) | 9 (10) | 28 (39)
Upper respiratory tract infection (Infections and infestations) | 16 (16) | 17 (20) | 8 (10)
Urinary tract infection (Infections and infestations) | 10 (11) | 11 (13) | 6 (7)
Decreased appetite (Metabolism and nutrition disorders) | 18 (22) | 12 (15) | 12 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 9 (11) | 12 (13)
Dizziness (Nervous system disorders) | 5 (6) | 12 (13) | 9 (12)
Headache (Nervous system disorders) | 10 (14) | 14 (57) | 20 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days